CLINICAL TRIAL: NCT02827526
Title: Methadone and Ketamine for Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH15-268
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2020-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Active Comparator): Patients in the ketamine arm will receive an intraoperative and postoperative infusion of ketamine
  Interventions: Drug: Ketamine
- Control (Placebo Comparator): Patients in the control arm will receive an intraoperative and postoperative infusion of dextrose
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Ketamine
  Arms: Ketamine
Drug: Control
  Other Names: dextrose infusion
  Arms: Control

SUMMARY:
Patients undergoing major spinal surgery continue to experience moderate-to-severe pain during the first 2-3 days following the operative procedure. Several factors contribute to postoperative pain in this patient population. Many patients present to surgery dependent on relatively high doses of oral opioids; this daily administration leads to tolerance to the effects of these drugs as well as hyperalgesia (exposure to opioids makes subsequent pain worse). In addition, surgical procedures on the spine are very painful. Furthermore, most of the opioids used after surgery only produce analgesia (pain relief) for 2-4 hours, which leads to fluctuations in levels of pain control (patients have to push a button to deliver pain medication when they begin to feel discomfort). Recent data suggest that the use of a long-acting opioid like methadone in the operating room, which provides analgesia for 24-36 hours, may improve pain control after spinal fusion surgery. However, other pain treatment modalities are required in this patient population. Studies have demonstrated that ketamine, a drug that prevents pain by a mechanism different from opioids, is effective in reducing pain medication requirements when given in the perioperative period. Small-dose infusions not only provide analgesia, but also prevent opioid tolerance and hyperalgesia. In particular, the combination of methadone and ketamine may be especially effective in controlling pain in patients following major operations. The aim of this randomized clinical trial is to examine the effect of a low-dose perioperative infusion of ketamine, when given with methadone in the operating room, on postoperative pain medication requirements, pain scores, and clinical recovery characteristics after spinal fusion surgery.

DETAILED DESCRIPTION:
Methadone is an opioid with the potential to provide prolonged and constant analgesia. It has a half-life that is significantly longer than other clinically-used opioids (25-52 hours). This unique property of methadone suggests that a single dose administered in the operating room can result in extended pain relief following surgery. When given intravenously to surgical patients, a half-life of 35 hours was observed, resulting in a median duration of analgesia of 26 hours. In patients undergoing abdominal, orthopedic, or gynecologic surgery, the use of a single dose of methadone (20 mg or 0.2-0.3 mg/kg) at induction of anesthesia resulted in reduced analgesic requirements and improved pain scores for the first 24-48 postoperative hours (when compared to patients given traditional intraoperative opioids). Only one retrospective study has examined the use of intraoperative methadone in adult patients undergoing spinal instrumentation. In this investigation, methadone use was associated with a 50% reduction in postoperative opioid requirements, compared to patients receiving shorter-acting opioids. Despite the use of methadone and postoperative PCA opioids, however, average pain scores were greater than 3 (on a 0 to 10 scale) in the methadone group. These findings suggest that methadone alone is insufficient in alleviating pain after major spine surgery.

A large number of clinical trials have examined the use of ketamine in the perioperative period. Several systematic reviews and meta-analyses have assessed the benefits and risks of ketamine in surgical patients. Bell et al. concluded that perioperative ketamine reduced analgesic requirements or pain intensity, or both. The incidence of nausea and vomiting was reduced, and adverse events were mild or absent. Himmelseher et al. noted that intravenous subanesthetic ketamine in general anesthesia provided pain prevention after surgery. Jouguelet-Lacoste et al. determined that low-dose ketamine reduced opioid consumption by 40%. Pain scores were also reduced, and no major complications were noted. Laskowski et al. concluded that ketamine resulted in a reduction in opioid consumption across all studies, and lower pain score were reported in most investigations. No significant differences in adverse events were noted in most meta-analyses, with the exception of a lower risk of nausea and vomiting in patients randomized to receive ketamine (a higher risk of hallucinations was reported in one meta-analysis). A large number of different dosing strategies have been used for ketamine. However, the greatest efficacy appears to result when a bolus dose is given (0.5 mg/kg) before incision, followed by an intraoperative (0.25-0.5 mg/kg/hr) infusion, and a postoperative (0.06-0.12 mg/kg/hr) infusion continued for at least 24-48 hours

Like methadone, ketamine is used most frequently in patients undergoing spinal fusion surgery due to the high incidence of pre-existing opioid tolerance and hyperalgesia (personal communication). Ketamine infusions have been investigated in 6 randomized studies in this patient population. In 5 of the trials, reduced postoperative opioid requirements, decreased pain scores, or both, were observed in patients randomized to receive ketamine. Shorter-acting opioids were used with ketamine in 5 of the investigations. Despite data suggesting a beneficial effect of ketamine in patients undergoing major spine surgery, a recent "best evidence" review stated that "there is insufficient and /or conflicting evidence that ketamine provides a significant reduction in postoperative pain or narcotic usage"

In theory, the use of a combination of a long-acting opioid and ketamine may be particularly efficacious in optimizing postoperative pain management. Recent evidence has demonstrated that methadone, like ketamine, has the ability to block NMDA receptors. In a neuropathic animal model, the combination of methadone and ketamine produced an analgesic synergy of a supra-additive nature. In the clinical setting, the administration of methadone and ketamine has only been examined in one small trial (20 patients). Patients randomized to receive methadone and ketamine required 70% less pain medication than those administered methadone alone. Although clinicians at NorthShore and other institutions are beginning to use methadone and ketamine in patients undergoing spinal surgery, there is limited evidence examining this approach in this patient population.

The primary aim of this randomized, double-blind study is to examine a perioperative analgesic strategy utilizing both ketamine and methadone in patients undergoing posterior spinal fusion. Patients randomized to the ketamine group will be given 0.2 mg/kg of methadone at anesthetic induction, and a ketamine infusion will be used intraoperatively and for 48 hours after surgery. Patients in the control group will receive 0.2 mg/kg of methadone at anesthetic induction, and then a D5W (sugar water) infusion intraoperatively and for 48 hours postoperatively. The total amount of PCA hydromorphone used postoperatively will be recorded, as well as postoperative pain scores. Recovery variables will be measured and patients will be assessed for adverse events potentially related to opioids and ketamine. NMDA receptor stimulation is also thought to play an important role in the development of chronic pain after surgery. Therefore, patients will be surveyed about chronic postsurgical pain 1, 3, 6, and 12 months after the operation to determine whether intraoperative management may influence the development of long-term adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for elective posterior spinal fusion surgery (lower thoracic, lumbar, sacral)
* Ages 18-80

Exclusion Criteria:

* Preoperative renal failure (defined as a serum creatinine > 2.0 mg/dL.)
* American Society of Anesthesiologists Physical Status IV or V
* Pulmonary disease necessitating home oxygen therapy
* Allergy to methadone, hydromorphone, or ketamine
* Preoperative recent history of opioid or alcohol abuse
* Significant liver disease
* Inability to use a PCA device or speak the English language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
hydromorphone consumption | first 24 hours

SECONDARY OUTCOMES:
hydromorphone consumption | second 24 hours
hydromorphone consumption | third 24 hours
postoperative pain | morning of postoperative day 1
  scale of 0 to 10 (0=no pain 10=worst pain imaginable))
postoperative pain | morning of postoperative day 2
  scale of 0 to 10, 0=no pain, 10=worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No